CLINICAL TRIAL: NCT02797964
Title: A Phase 1/2 Trial of SRA737 (a Chk1 Inhibitor) Administered Orally in Subjects With Advanced Cancer
Brief Title: A Phase 1/2 Trial of SRA737 in Subjects With Advanced Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sierra Oncology LLC - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SRA737-01
Record Dates: First submitted 2016-05-23; First posted 2016-06-14 (Estimated); Results first posted 2022-03-10 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Advanced Solid Tumors or Non-Hodgkin's Lymphoma (NHL)
Keywords: Replication stress; Advanced solid tumors; CCNE1; TP53; BRCA1; BRCA2; MYC; RAD50; Fanconi anemia; Cell cycle; Metastatic Colorectal Cancer; Platinum-Resistant or Intolerant High Grade Serious Ovarian Cancer; Advanced Non-Small Cell Lung Cancer; Metastatic Castration-Resistant Prostate Cancer; Head and Neck Squamous Cell Carcinoma; Squamous Cell Carcinoma of the Anus; Phase 1; Phase 2; Dose escalation; Chk1 inhibitor; Checkpoint kinase 1; Synthetic lethality; Next-Generation Sequencing; Genetic biomarkers
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Fanconi Anemia; Colorectal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Anus Neoplasms | interventions — SRA737

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label (Experimental)
  Interventions: Drug: SRA737

INTERVENTIONS:
Drug: SRA737 — SRA737 will be administered orally on each day of a 28-day cycle. Subjects will receive a single dose of SRA737 between 4 to 7 days prior to starting the first cycle for PK profiling. Subjects can continue taking SRA737 if they are receiving clinical benefit and able to safely take the drug and follow the requirements of the study.

SUMMARY:
The purpose of this clinical study is to establish the safety profile, determine the maximum tolerated dose (MTD) and recommend a Phase 2 dose and schedule of SRA737; and to evaluate the efficacy of SRA737 in prospectively-selected subjects with genetically-defined tumors that harbor genomic alterations linked to increased replication stress and that are hypothesized to be more sensitive to checkpoint kinase 1 (Chk1) inhibition via synthetic lethality. Specific cancer indications that frequently harbor these genetic mutations will be studied.

DETAILED DESCRIPTION:
SRA737 is a potent, highly selective, orally bioavailable small molecule inhibitor of Chk1, a key regulator of cell cycle progression and the DNA Damage Response (DDR) replication stress response. In cancer cells, intrinsic replication stress (RS) is induced by factors such as oncogenes (e.g., CCNE1 or MYC), genetic mutations in DNA repair machinery (e.g. BRCA1 or FANCA), genetic mutations leading to a dysregulated cell cycle (e.g., TP53 or RAD50) or other genomic alterations. This replication stress results in persistent DNA damage and genomic instability, leading to an increased dependency on Chk1 for survival. Targeted inhibition of Chk1 by SRA737 may therefore be synthetically lethal to cancer cells with elevated intrinsic RS.

This study has been designed to: establish the safety profile; determine the pharmacokinetic profile; identify the optimal dose, schedule, and MTD; obtain preliminary evidence of activity; and evaluate SRA737's efficacy in prospectively-selected subjects with tumors that harbor genomic alterations linked to increased replication stress and that are hypothesized to be more sensitive to Chk1 inhibition via synthetic lethality.

This clinical study consists of two phases, a Dose Escalation Phase 1 portion and a Cohort Expansion Phase 2 portion.

In the Dose Escalation Phase 1 portion, cohorts consisting initially of a single subject will receive escalating doses of SRA737, administered orally on a continuous daily dosing schedule in 28-day cycles. Once an SRA737-related Grade 2 toxicity is observed in a dose escalation cohort during Cycle 1, that cohort will be expanded to 3 to 6 subjects, and subsequent dose level cohorts will follow a rolling 6 design until the MTD has been identified.

In the Cohort Expansion Phase 2 portion, subjects with genetically-defined tumors that harbor genomic alterations linked to increased replication stress and that are hypothesized to be more sensitive to Chk1 inhibition will be prospectively enrolled into six indication-specific cohorts to explore the preliminary efficacy of SRA737. Subjects must have advanced or metastatic disease of one of the following types:

* castration-resistant prostate cancer (mCRPC);
* high grade serous ovarian cancer (HGSOC) without CCNE1 gene amplification;
* HGSOC with CCNE1 gene amplification (or alternative genetic alteration with similar functional effect);
* non-small cell lung cancer (NSCLC);
* head and neck squamous cell carcinoma (HNSCC) or squamous cell carcinoma of the anus (SCCA); and
* colorectal cancer (mCRC).

To qualify for enrolment in the Cohort Expansion Phase 2 portion, the subject's tumor must have a confirmed combination of mutations which are expected to confer sensitivity to Chk1 inhibition, determined by the Sponsor's review of genetic abnormalities detected in the following categories:

* Oncogenic drivers such as CCNE1 or MYC, etc.
* Genes involved in the DNA repair process including BRCA1, BRCA2, FANC genes, mismatch repair (MMR) genetic alterations and/or high microsatellite instability.
* Key tumor suppressor genes regulating G1 cell cycle progression/arrest such as TP53, RAD50, etc. For patients with HNSCC or SCCA, positive human papilloma virus (HPV) status is also considered for eligibility.
* Genetic indicators of replicative stress such as gain of function/amplification of CHEK1, ATR or other related genes.

Tumor genetics will be prospectively determined using Next-Generation Sequencing.

ELIGIBILITY:
Key Inclusion Criteria:

1. For Dose Escalation Only: any locally advanced or metastatic, histologically or cytologically proven solid tumor or NHL, relapsed after or progressing despite conventional treatment
2. Life expectancy of at least 12 weeks
3. World Health Organization (WHO) performance status of 0-1
4. Must meet select hematological and biochemical laboratory indices
5. Archival tumor tissue or accessible tumor and willingness to consent to a biopsy

Expansion Only:

1. Any locally advanced or metastatic malignancy of the following types for which no other conventional therapy is considered appropriate:

   * Metastatic Colorectal Cancer (CRC)
   * Platinum-resistant or intolerant High Grade Serious Ovarian Cancer (HGSOC)
   * Advanced Non-Small Cell Lung Cancer (NSCLC)
   * Metastatic Castration-Resistant Prostate Cancer (mCRPC)
   * Head and Neck Squamous Cell Carcinoma (HNSCC) or squamous cell carcinoma of the anus (SCCA).
   * Eligibility may be further restricted by the select number of prior regimens specific to each indication
2. Measurable disease per RECIST v1.1, or for mCRPC, evaluable disease per any of the following:

   * Measurable disease per RECIST v1.1
   * Increasing PSA
   * Circulating tumor cell (CTC) count of 5 or more cells per 7.5 ml of blood
3. Tumor tissue or ctDNA evidence that subject's tumor harbors a combination of mutations which are expected to confer sensitivity to Chk1 inhibition. Eligibility will be determined by the Sponsor's review of genetic abnormalities detected in genes in the following categories:

   * Oncogenic drivers such as MYC, CCNE1, etc.
   * Key tumor suppressor genes regulating G1 cell cycle progression/arrest such as RAD50, TP53, etc. For patients with NHSCC or SCCA, positive HPV status is also considered for eligibility.
   * The DDR pathway including BRCA1, BRCA2 and FANC. For patients with CRC, MMR genetic alterations and/or high microsatellite instability are also considered for eligibility.
   * Genetic indicators of replicative stress such as gain of function/amplification of Chk1 or ATR or other related gene.

Key Exclusion Criteria:

1. Received the following prior or current anticancer therapy:

   * Radiotherapy within the last 6 weeks
   * Endocrine therapy during the previous 4 weeks
   * Chemotherapy during the previous 4 weeks
   * Immunotherapy during the previous 6 weeks
   * Nitrosoureas or Mitomycin C during the previous 6 weeks
   * Other Investigational Medicinal Product during the 4 weeks before treatment
   * Any prior treatment with a Chk1 inhibitor or prior treatment with an ATR inhibitor within 6 months prior to receiving SRA737
2. Other malignancy within the past 2 years, except for adequately treated tumors
3. Ongoing toxic manifestations of previous treatments greater than NCI-CTCAE Grade 1
4. For Dose Escalation: new or progressing brain metastases. For Cohort Expansion: present or prior brain metastases
5. High medical risk because of nonmalignant systemic disease
6. Serologically positive for hepatitis B, hepatitis C or HIV
7. Serious cardiac condition, left ventricular ejection fraction < 45% at baseline, history of cardiac ischemia within the past 6 months, or prior history of cardiac arrhythmia requiring treatment
8. Prior bone marrow transplant or extensive radiotherapy to greater than 25% of bone marrow within 8 weeks
9. Peanut allergy
10. QTcF> 450 msec in adult males and > 470 msec in adult females
11. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of SRA737
12. Inability to swallow capsules without chewing or crushing
13. Is a participant or plans to participate in another interventional clinical trial
14. Any other condition which in the Investigator's opinion would not make the subject a good candidate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2019-10-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United Kingdom (15):
  - Royal Marsden Hospital, Sutton, London
  - Belfast City Hospital, Belfast, Northern Ireland
  - Oxford University Hospitals, Headington, Oxford
  - Velindre Cancer Centre - Cardiff, Cardiff, Whitchurch
  - The Clatterbridge Cancer Centre, Bebington, Wirral
  - Western General Hospital, Edinburgh
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - The Leeds Teaching Hospitals of St James University Hospital, Leeds
  - University Hospitals of Leicester, Leicester
  - Guy's and St. Thomas, London
  - Sarah Cannon Research Institute, London
  - University College London Hospitals, London
  - The Christie, Manchester
  - Freeman Hospital, Newcastle upon Tyne
  - Sheffield Teaching Hospitals, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kristeleit R, Plummer R, Jones R, Carter L, Blagden S, Sarker D, Arkenau T, Evans TRJ, Danson S, Symeonides SN, Veal GJ, Klencke BJ, Kowalski MM, Banerji U. A Phase 1/2 trial of SRA737 (a Chk1 inhibitor) administered orally in patients with advanced cancer. Br J Cancer. 2023 Jul;129(1):38-45. doi: 10.1038/s41416-023-02279-x. Epub 2023 Apr 29. PMID 37120671
- [Derived] Jin T, Xu L, Wang P, Hu X, Zhang R, Wu Z, Du W, Kan W, Li K, Wang C, Zhou Y, Li J, Liu T. Discovery and Development of a Potent, Selective, and Orally Bioavailable CHK1 Inhibitor Candidate: 5-((4-((3-Amino-3-methylbutyl)amino)-5-(trifluoromethyl)pyrimidin-2-yl)amino)picolinonitrile. J Med Chem. 2021 Oct 28;64(20):15069-15090. doi: 10.1021/acs.jmedchem.1c00994. Epub 2021 Oct 19. PMID 34665631

RESULTS

PARTICIPANT FLOW:
Groups:
- Colorectal Cancer: Metastatic colorectal cancer (CRC) defined as histologically and/or cytologically confirmed CRC, and must have received at least 1 prior regimen for advanced/metastatic disease.
- High Grade Serous Ovarian Cancer: High grade serous ovarian cancer (HGSOC) defined as histologically confirmed high grade serous ovarian, fallopian tube or primary peritoneal cancer who were recurrent platinum intolerant, or with platinum resistant disease defined as radiological evidence of disease progression within 6 months of the last receipt of platinum based chemotherapy.
- Non Small Cell Lung Cancer: Advanced non small cell lung cancer (NSCLC) defined as locally advanced and recurrent or metastatic, histologically confirmed NSCLC, and must have received at least 1 prior regimen for advanced/metastatic disease.
- Metastatic Other Tumor Type Castration Resistant Prostate Cancer: Metastatic castration resistant prostate cancer (mCRPC) defined as histologically or cytologically confirmed adenocarcinoma of the prostate that has progressed after androgen deprivation therapy.
- Head and Neck Squamous Cell Carcinoma: Histologically confirmed HNSCC from any primary site; locally advanced disease (ie, persistent or progressive disease following curative intent radiation, and not a candidate for surgical salvage due to incurability or morbidity), or metastatic disease.
- Other Tumor Type: Any locally advanced or metastatic, histologically or cytologically proven solid tumor or NHL, that had relapsed after or progressing despite conventional treatment for which no conventional therapy was considered appropriate by the investigator or had been declined by the subject.
Period: Overall Study
Arm/Group | Colorectal Cancer | High Grade Serous Ovarian Cancer | Non Small Cell Lung Cancer | Metastatic Other Tumor Type Castration Resistant Prostate Cancer | Head and Neck Squamous Cell Carcinoma | Other Tumor Type
Started | 32 | 37 | 10 | 16 | 4 | 8
Completed | 32 | 37 | 10 | 16 | 4 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Evaluable Population includes all enrolled subjects who receive at least 1 dose of SRA737.
Groups:
- Total: Total of all reporting groups
Arm/Group | Colorectal Cancer | High Grade Serous Ovarian Cancer | Non Small Cell Lung Cancer | Metastatic Other Tumor Type Castration Resistant Prostate Cancer | Head and Neck Squamous Cell Carcinoma | Other Tumor Type | Total
Number analyzed (Participants) | 32 | 37 | 10 | 16 | 4 | 8 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (12.05) | 60.6 (9.81) | 64.4 (9.11) | 68.3 (6.76) | 63.0 (6.06) | 58.4 (6.46) | 62.2 (10.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 37 | 6 | 0 | 0 | 4 | 61
  Male | 18 | 0 | 4 | 16 | 4 | 4 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 30 | 32 | 10 | 15 | 4 | 8 | 99
  Unknown or Not Reported | 2 | 5 | 0 | 1 | 0 | 0 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 0 | 0 | 2
  Black or African American | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 29 | 35 | 10 | 13 | 4 | 8 | 99
  Other | 2 | 2 | 0 | 0 | 0 | 0 | 4
  Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 32 | 37 | 10 | 16 | 4 | 8 | 107

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events as Assessed by CTCAE 4.03
Description: Treatment-emergent adverse events (TEAEs) were reported until the safety Follow up (SFU) visit, 30 days after the last dose of SRA737 or prior to the initiation of a new anticancer treatment, whichever came first.
Time Frame: Up to 30 days after last dose of SRA737
Population: As specified in the Statistical Analysis Plan, the frequency of each AE was evaluated in the overall Safety Evaluable Population rather than by tumor type subgroups with the intention of displaying the overall safety profile of SRA737 in advanced solid tumors. The Safety Evaluable Population includes all enrolled subjects who receive at least 1 dose of SRA737.
Measure: Count of Participants; unit: Participants
Groups:
- Safety Evaluable Population: The Safety Evaluable Population includes all enrolled subjects who receive at least 1 dose of SRA737.
Arm/Group | Safety Evaluable Population
Number analyzed (Participants) | 107
Participants | 106

2. Primary Outcome: Maximum Tolerated Dose of SRA737
Description: The highest dose at which ≤ 33% of subjects have a dose limiting toxicity (DLT) in a cohort of up to 6 subjects.
Time Frame: Cycle 1 (28 days) in the Dose Escalation Phase
Population: In order to determine the MTD, a total of 18 subjects were enrolled in the dose escalation phase of the study in 9 dosage cohorts. All subjects receiving at least 75% of planned doses of SRA737 within Cycle 1 and those subjects receiving less than these planned doses of SRA737 due to DLT were considered evaluable for dose review decisions.
Measure: Number; unit: mg QD
Groups:
- Dose Escalation Phase: The Dose Escalation Phase included a total of 18 subjects in 9 different dosage cohorts: 20 mg QD, 40 mg QD, 80 mg QD, 160 mg QD, 300 mg QD, 600 mg QD, 1000 mg QD, 500 mg BID, and 1300 mg QD.
Arm/Group | Dose Escalation Phase
Number analyzed (Participants) | 18
mg QD | 1000

3. Primary Outcome: Recommended Phase 2 Dose of SRA737
Description: The RP2D and schedule were defined by the Cohort Review Committee at the end of the study and took all clinically relevant toxicity, PK and PDn data into account. The RP2D was to be a dose equal to or less than the MTD for the selected schedule.
Time Frame: Up to 30 days after last dose of SRA737
Population: All 107 subjects treated in the study were included in the review of toxicity, PK and PDn, data in order to determine the RP2D. All clinically relevant toxicity, PK and PDn data up to 30 days after last dose of SRA737 were taken into account.
Measure: Number; unit: mg QD
Arm/Group | Safety Evaluable Population
Number analyzed (Participants) | 107
mg QD | 800

4. Primary Outcome: Disease Control Rate (DCR) of SRA737
Description: The disease control rate (DCR) was defined as the number of subjects achieving complete response (CR) + partial response (PR) + stable disease (SD) per RECIST 1.1 criteria. Since no subjects achieved CR or PR in this study, the DCR represents the proportion of subjects in each group who achieved SD.
Time Frame: Radiographic tumor assessments were performed every 2 cycles of therapy.
Population: The Response Evaluable Population (REP) included all enrolled subjects who satisfy all of the following conditions:
  1. Measurable disease and assessment at baseline
  2. Received at least 75% of 1 cycle of study medication, based on dosing information
  3. At least one post baseline disease assessment OR discontinued treatment due to AE or disease progression or death
Measure: Count of Participants; unit: Participants
Arm/Group | Colorectal Cancer | High Grade Serous Ovarian Cancer | Non Small Cell Lung Cancer | Metastatic Other Tumor Type Castration Resistant Prostate Cancer | Head and Neck Squamous Cell Carcinoma
Number analyzed (Participants) | 25 | 26 | 8 | 13 | 4
Participants | 8 | 11 | 3 | 8 | 3

5. Primary Outcome: Time to Progression (TTP)
Description: Time to progression (TTP) was defined as the time from Cycle 1 Day 1 to the earliest date of radiographic disease progression per RECIST 1.1, or if the subject did not experience disease progression, to the last imaging assessment. TTP was analyzed using the K-M method.
Time Frame: Radiographic tumor assessments were performed every 2 cycles of therapy. Follow-up assessments were made every 16 weeks for subjects who had not progressed and had not initiated new anticancer therapy.
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Colorectal Cancer | High Grade Serous Ovarian Cancer | Non Small Cell Lung Cancer | Metastatic Other Tumor Type Castration Resistant Prostate Cancer | Head and Neck Squamous Cell Carcinoma
Number analyzed (Participants) | 24 | 26 | 8 | 13 | 4
months | 1.87 [1.68 to 3.06] | 1.94 [1.81 to 3.68] | 1.87 [1.41 to NA] — The upper 95% CI was not estimated due to insufficient number of participants with events | 3.02 [1.64 to NA] — The upper 95% CI was not estimated due to insufficient number of participants with events | 3.87 [1.64 to NA] — The upper 95% CI was not estimated due to insufficient number of participants with events

6. Primary Outcome: Progression Free Survival (PFS)
Description: Progression free survival (PFS) was defined as time from Cycle 1 Day 1 to the earliest date of radiographic disease progression per RECIST 1.1 or death, whichever happened first. Censoring rules are defined in the SAP. PFS was analyzed using the K-M method.
Time Frame: as for outcome 5
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Colorectal Cancer | High Grade Serous Ovarian Cancer | Non Small Cell Lung Cancer | Metastatic Other Tumor Type Castration Resistant Prostate Cancer | Head and Neck Squamous Cell Carcinoma
Number analyzed (Participants) | 24 | 26 | 8 | 13 | 4
months | 1.84 [1.68 to 1.87] | 1.94 [1.81 to 3.68] | 1.76 [0.49 to NA] — The upper 95% CI was not estimated due to insufficient number of participants with events | 3.02 [1.64 to NA] — The upper 95% CI was not estimated due to insufficient number of participants with events | 3.55 [1.64 to NA] — The upper 95% CI was not estimated due to insufficient number of participants with events

7. Primary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was defined as time from Cycle 1 Day 1 to the date of death (or date last known to be alive). OS was analyzed using the K-M method.
Time Frame: Follow-up assessments were made every 16 weeks for subjects who had not progressed and had not initiated new anticancer therapy.
Population: The Response Evaluable Population (REP) included all subjects who satisfy the following conditions:
  1. Measurable disease and assessment at baseline
  2. Received at least 75% of 1 cycle of study medication, based on dosing information
  3. At least 1 post baseline disease assessment OR discontinued treatment due to AE or disease progression or death Note: The median OS was not estimated in the mCRPC, HNSCC, or "Other" tumor type subgroups due to insufficient number of participants with events.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Metastatic Castration Resistant Prostate Cancer: Metastatic castration resistant prostate cancer (mCRPC) defined as histologically or cytologically confirmed adenocarcinoma of the prostate that has progressed after androgen deprivation therapy.
- Overall: All subjects included in the Response Evaluable Population
Arm/Group | Colorectal Cancer | High Grade Serous Ovarian Cancer | Non Small Cell Lung Cancer | Metastatic Castration Resistant Prostate Cancer | Head and Neck Squamous Cell Carcinoma | Other Tumor Type | Overall
Number analyzed (Participants) | 24 | 26 | 8 | 13 | 4 | 8 | 81
months | 5.72 [4.14 to NA] — The upper 95% CI was not estimated due to insufficient number of participants with events | 6.93 [4.80 to NA] — The upper 95% CI was not estimated due to insufficient number of participants with events | 6.08 [0.49 to NA] — The upper 95% CI was not estimated due to insufficient number of participants with events | NA [NA to NA] — The median and 95% CIs were not estimated due to insufficient number of participants with events | NA [3.55 to NA] — The median and upper 95% CI were not estimated due to insufficient number of participants with events | NA [1.64 to NA] — The median and upper 95% CI were not estimated due to insufficient number of participants with events | 6.93 [5.72 to NA] — The upper 95% CI was not estimated due to insufficient number of participants with events

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were reported until the safety Follow up (SFU) visit, 30 days after the last dose of SRA737 or prior to the initiation of a new anticancer treatment, whichever came first. Long term Follow up (LTFU) visits were conducted every 16 weeks for subjects who had not progressed and had not initiated new anticancer therapy.
Description: An AE was defined as any untoward, undesired, or unplanned medical occurrence in a subject administered SRA737. All AEs and SAEs were assessed for seriousness, causality, and expectedness.
  As specified in the Statistical Analysis Plan, the frequency of each AE was evaluated in the overall Safety Evaluable Population (all enrolled subjects who receive at least 1 dose of SRA737) of patients with advanced solid tumors, irrespective of tumor type. All AEs collected are included in the summary.
Groups:
- Safety Evaluable Population: Due to the small numbers of patients in some tumor type subgroups and with the intention of displaying the overall safety profile of SRA737 in advanced solid tumors, the frequency of each AE was evaluated in the overall Safety Evaluable Population rather than by tumor type subgroups. The Safety Evaluable Population includes all enrolled subjects who receive at least 1 dose of SRA737.
Arm/Group | Safety Evaluable Population
All-Cause Mortality (participants affected / at risk) | 18/107
Serious Adverse Events (participants affected / at risk) | 48/107
Other Adverse Events (participants affected / at risk) | 106/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Evaluable Population (N=107)
Disease progression (General disorders) | 10 (10)
Pyrexia (General disorders) | 4 (4)
Infection (Infections and infestations) | 4 (4)
Lung infection (Infections and infestations) | 2 (2)
Abdominal sepsis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Intestinal sepsis (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (2)
Lymphangitis (Infections and infestations) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 2 (2)
Biopsy liver (Investigations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
Spinal cord compression (Musculoskeletal and connective tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Evaluable Population (N=107)
Diarrhoea (Gastrointestinal disorders) | 74 (131)
Nausea (Gastrointestinal disorders) | 72 (125)
Vomiting (Gastrointestinal disorders) | 56 (94)
Constipation (Gastrointestinal disorders) | 19 (26)
Abdominal pain (Gastrointestinal disorders) | 17 (23)
Abdominal distension (Gastrointestinal disorders) | 11 (17)
Dyspepsia (Gastrointestinal disorders) | 10 (11)
Abdominal pain upper (Gastrointestinal disorders) | 7 (7)
Ascites (Gastrointestinal disorders) | 6 (7)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (6)
Fatigue (General disorders) | 54 (85)
Pyrexia (General disorders) | 13 (13)
Decreased appetite (Metabolism and nutrition disorders) | 26 (36)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (9)
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 (9)
Hyponatraemia (Metabolism and nutrition disorders) | 8 (21)
Headache (Nervous system disorders) | 13 (13)
Lethargy (Nervous system disorders) | 9 (14)
Dysgeusia (Nervous system disorders) | 8 (9)
Dizziness (Nervous system disorders) | 7 (7)
Urinary tract infection (Infections and infestations) | 12 (15)
Oral candidiasis (Infections and infestations) | 7 (7)
Cellulitis (Infections and infestations) | 6 (8)
Lower respiratory tract infection (Infections and infestations) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 6 (8)
Blood alkaline phosphatase increased (Investigations) | 18 (22)
Aspartate aminotransferase increased (Investigations) | 14 (21)
Alanine aminotransferase increased (Investigations) | 11 (19)
Lymphocyte count decreased (Investigations) | 10 (32)
Blood creatinine increased (Investigations) | 7 (9)
Electrocardiogram QT prolonged (Investigations) | 7 (10)
White blood cell count decreased (Investigations) | 7 (24)
Gamma-glutamyltransferase increased (Investigations) | 6 (6)
Platelet count decreased (Investigations) | 6 (14)
Anaemia (Blood and lymphatic system disorders) | 25 (48)
Neutropenia (Blood and lymphatic system disorders) | 16 (34)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (16)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 (23)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (11)
Rash (Skin and subcutaneous tissue disorders) | 11 (18)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8)
Hypotension (Vascular disorders) | 6 (7)
Insomnia (Psychiatric disorders) | 8 (9)
Tachycardia (Cardiac disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All proposed publications and presentations by the investigators, personnel, or associates resulting from or relating to this study must be submitted to Sierra Oncology for review before submission for publication or presentation. If the proposed publication or presentation contains patentable subject matter, which, at Sierra Oncology's sole discretion, warrants intellectual property protection, Sierra Oncology may delay publication or presentation for the purpose of pursuing such protection.

DOCUMENTS (2):
  • Study Protocol (2018-01-10): https://cdn.clinicaltrials.gov/large-docs/64/NCT02797964/Prot_000.pdf
  • Statistical Analysis Plan: Revised (final) statistical analyses (2021-01-22): https://cdn.clinicaltrials.gov/large-docs/64/NCT02797964/SAP_001.pdf